CLINICAL TRIAL: NCT04728516
Title: The Effect of Vonoprazan-based Dual Eradication Therapy vs PPI Treatment on Gastrointestinal Bleeding in ACS Patients With Hp Infection and Coronary Stents: an Open-label, Randomized, Controlled Trial
Brief Title: The Effect of Dual Eradication Therapy vs PPI on Gastrointestinal Bleeding in ACS Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020SDUCRCA006
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome; Helicobacter Pylori Infection
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Amoxicillin; Pantoprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan-based dual eradication therapy (Experimental): H. pylori eradication using a dual eradication regimen, a course of 14 days, followed up to 6 months after randomization; the treatment regimen is as follows: routine use of Vonoprazan 20mg bid + amoxicillin 1g tid, a course of 14 days .
  Interventions: Drug: Vonoprazan-based dual eradication therapy for two weeks; Drug: amoxicillin
- Pantoprazole (Active Comparator): To take pantoprazole 40 mg daily, followed up to 6 months after randomization.
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Vonoprazan-based dual eradication therapy for two weeks — Patients with ACS after PCI, associated with positive Hp need a long-term DAPT treatment. We conducted a study on the prevention of gastrointestinal bleeding between vonoprazan-based dual eradication therapy for two weeks and pantoprazole for six months of a rountine therapy.
  Arms: Vonoprazan-based dual eradication therapy
Drug: amoxicillin — amoxicillin
  Arms: Vonoprazan-based dual eradication therapy
Drug: Pantoprazole — Pantoprazole
  Arms: Pantoprazole

SUMMARY:
Patients with acute coronary syndrome (ACS) after Percutaneous Coronary Intervention (PCI) require routine treatment with dual antiplatelet (DAPT) treatment, but with the high risk of bleeding, gastrointestinal bleeding is the most common type of major bleeding. Helicobacter pylori (Hp) infection is a high-risk factor for gastrointestinal bleeding, with an incidence of about 50%. Foreign authoritative DAPT guidelines do not give individual guidance to Hp-infected patients. It is recommended that those with high bleeding risk should be combined with proton pump inhibitors (PPI), but long-term compliance with PPI is not ideal. Authoritative experts in China have agreed to recommend Hp detection and eradication therapy for DAPT patients, but loss of evidence. Vonoprazan is a novel potassium ion competitive acid blocker, based on Vonoprazan's dual Hp eradication therapy is simple and effective. Our team will conduct a multi-center, open-label, randomized controlled clinical trial using a non-inferior design to compare the combination of Vonoprazan + amoxicillin combined with pantoprazole (PPI) for 6 months after PCI on the bleeding events of the digestive tract.

DETAILED DESCRIPTION:
This study plans to enroll 2600 patients, 1300 patients in each group, in the project participating hospitals who received coronary stenting and are expected to undergo DAPT ≥6 months after operation. Hp13C-urea breath test and serum Hp antibody scores Type detection, patients with positive Hp infection.

Antiplatelet drugs (DAPT) use aspirin 100 mg qd, plus clopidogrel 75 mg qd or aspirin 100mg qd plus ticagrelor 90 mg bid. The specific medication is evaluated and decided by the interventional doctor.

After the subjects in each center signed a written informed consent form, they randomly divided each test case into a test group or a control group at a 1:1 ratio:

1. Test group:

   In the project participating hospitals who received coronary stenting and are expected to undergo DAPT ≥6 months after operation. Hp13C-urea breath test and serum Hp antibody scores Type detection, patients with positive Hp infection. Antiplatelet drugs (DAPT) use aspirin 100 mg qd, plus clopidogrel 75 mg qd or aspirin 100 mg qd, plus ticagrelor 90 mg bid. The specific medication is evaluated and decided by the interventional doctor.

   H. pylori eradication using a dual eradication regimen, a course of 14 days, followed up to 6 months after randomization; the treatment regimen is as follows: routine use of Vonoprazan 20mg bid + amoxicillin 1g tid, a duration of 14 days(Considering the high drug resistance rate of Hp strains in China, we increase the course of eradication treatment to 14 days) .

   i. Introduce the subject to the possible adverse reactions to the dual eradication at the informed stage, and inform the subject that when the adverse reaction occurs, the researcher should be contacted as soon as possible to deal with it as soon as possible to reduce unnecessary shedding. For patients who are unable to tolerate the combination therapy and fall off, record the reason for the incomplete treatment and the corresponding time point, and continue the safety visit.

   ii. More than 1 month after completion of the dual eradication (scheduled at the 12th week of follow-up, visit 3), use the 13C-urea breath test to retest Hp infection. For subjects who failed H. pylori eradication, in the Department of Gastroenterology Remedial treatment under the guidance of a doctor.
2. Control group:

In the project participating hospitals who received coronary stenting and are expected to undergo DAPT ≥ 6 months after operation. Hp13C-urea breath test and serum Hp antibody scores Type detection, patients with positive Hp infection. Antiplatelet drugs (DAPT) use aspirin 100 mg qd, plus clopidogrel 75 mg qd or aspirin 100 mg qd plus ticagrelor 90 mg bid. The specific medication is evaluated and decided by the interventional doctor. Taking pantoprazole 40 mg daily, followed up to 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACS and PCI treatment and postoperative DAPT ≥ 6 months;
2. Hp infection is positive;
3. Age ≥18 years old;
4. The patient himself or his authorized client signs the subject's consent.

Exclusion Criteria:

1. Previous history of gastrointestinal ulcer bleeding;
2. Long-term use of PPI and H2 receptor inhibitors in the past;
3. Complicated with gastroesophageal varices, or after gastrectomy;
4. Those who are taking anti-coagulation drugs such as vitamin K antagonists (warfarin) ,factor X or factor II inhibitors;
5. Recently received fibrinolytic therapy (using fibrin-specific drugs within 24 hours before randomization, or using non-fibrin-specific drugs within 48 hours before randomization);
6. Recently accepted (within 30 days before randomization) or planned to undergo coronary artery bypass grafting (CABG);
7. Combining active bleeding or coagulation dysfunction (indicator);
8. In patients with liver and kidney disease, serum creatinine is greater than 150 μmol/L, GFR <60ml/min/1.73m2, alanine aminotransferase and aspartate aminotransferase increase ≥3 times from the normal value;
9. Complicated with hemorrhagic stroke, intracranial tumor, arteriovenous malformation or aneurysm;
10. Anemia (adult male hemoglobin less than 120 g/L or red blood cells less than 4×10^12/L,adult female hemoglobin less than 105 g/L or red blood cells less than 3.5×10^12/L);
11. Systemic glucocorticoid application;
12. Have taken antibiotics and other drugs that affect the flora in the stomach within the past month;
13. A history of allergy to aspirin, clopidogrel, ticagrelor, pantoprazole, penicillin and other test drugs;
14. Pregnancy or breastfeeding women and subjects of childbearing age who do not want to take contraceptive measures;
15. With malignant tumors and other diseases, the expected survival time is less than 1 year;
16. Patients who participated in clinical trials of other drugs or are participating in clinical studies of other new drugs within 30 days before enrollment;
17. Complicated with mental illness or severe neurosis;
18. Can't express subjective discomfort symptoms;
19. The investigator decides that it is not suitable to participate in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal bleeding of 6 months in patients with ACS after PCI | 6 months
  To compare the effects of the combination of vonoprazan + amoxicillin and pantoprazole on gastrointestinal bleeding events within 6 months in patients with ACS after PCI，The primary endpoint was gastrointestinal bleeding, including gastroduodenal bleeding, gastrointestinal bleeding with unknown bleeding site, and occult gastrointestinal bleeding.

SECONDARY OUTCOMES:
major adverse cardiovascular and cerebrovascular events (MACCE) | 6 month
  To compare the effects of the combination of vonoprazan + amoxicillin and pantoprazole on major adverse cardiovascular and cerebrovascular events (MACCE) within 6 months in patients with ACS after PCI. The secondary outcomes measure were MACCE , including :stent thrombosis, recurrent myocardial infarction, unplanned revascularization cardiogenic shock, stroke, cardiovascular death, and all-cause death.
complex gastrointestinal event | 6month
  To compare the effects of the combination of vonoprazan + amoxicillin and pantoprazole on complex gastrointestinal events. The secondary outcomes measure were complex gastrointestinal events, including upper gastrointestinal bleeding (BARC type), symptomatic gastroduodenal ulcer, gastroesophageal reflux, intestinal obstruction, gastrointestinal perforation, diarrhea, dyspepsia.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-guo Chen, MD, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (42):
- China (42):
  - Bozhou People's Hospital, Bozhou, Anhui
  - Chuzhou First People's Hospital, Chuzhou, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Aviation General Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First People'S Hospital of Zunyi, Zunyi, Guizhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Qinghai Red Cross Hospital, Xining, Qinghai
  - Qilu Hospital of Shandong University Dezhou Hospital, Dezhou, Shandong
  - Pingyuan First People'S Hospital, Dezhou, Shandong
  - NINGJIN People's Hospital, Dezhou, Shandong
  - Dongying People's Hospital, Dongying, Shandong
  - THE Second People's Hospital of Dongying, Dongying, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - The 960th Hospital of the Joint Logistic Support Force, Jinan, Shandong
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - The fourth People's Hospital of jinan, Jinan, Shandong
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - JINA CITY People's Hospital, Jinan, Shandong
  - Central Hospital Affiliated to Shandong First medical University, Jinan, Shandong
  - The First People's Hospital of Jining City, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi City People's Hospital, Linyi, Shandong
  - Linshu County People'S Hospital, Linyi, Shandong
  - Qilu Hospital of Shandong University (Qingdao), Qingdao, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Weihai Central Hospital, Weihai, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Haiyang People's Hospital, Yantai, Shandong
  - Shandong Healthcare Group Zaozhuang Central Hospital, Zaozhuang, Shandong
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - The Ninth People's Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Ru Shan People's Hospital, Rushan, Yantai